CLINICAL TRIAL: NCT00794508
Title: MND-ADA Transduction of CD34+ Cells From the Bone Marrow Of Children With Adenosine Deaminase (ADA)-Deficient Severe Combined Immunodeficiency (SCID): Effect of Discontinuation of PEG-ADA and Marrow Cytoreduction With Busulfan
Brief Title: MND-ADA Transduction of CD34+ Cells From Children With ADA-SCID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Donald B. Kohn, M.D. (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Donald B. Kohn, M.D., Professor, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADA Gene Therapy; 1R01FD003005-01 (FDA); 9908-337 (Other: OBA-RAC)
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Severe Combined Immunodeficiency
Keywords: Severe Combined Immune Deficiency; Adenosine Deaminase Deficiency; Gene Therapy; Hematopoietic Stem Cells; Retroviral Vector; ADA-deficient SCID
MeSH Terms: conditions — Severe Combined Immunodeficiency; Severe combined immunodeficiency due to adenosine deaminase deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Retroviral-mediated ADA gene transfer (Experimental): Transfer of the human ADA gene to isolated CD34+ cells from the bone marrow.
  Interventions: Biological: ADA gene transfer

INTERVENTIONS:
Biological: ADA gene transfer — Autologous CD34+ cells transduced with the retroviral vector MND-ADA, carrying the human ADA gene.

SUMMARY:
Severe combined immune deficiency (SCID) may result from inherited deficiency of the enzyme adenosine deaminase (ADA). Children with ADA-deficient SCID often die from infections in infancy, unless treated with either a bone marrow transplant or with ongoing injections of PEG-ADA (Adagen) enzyme replacement therapy. Successful BMT requires the availability of a matched sibling donor for greatest success, and treatment using bone marrow from a less-well matched donor may have a higher rate of complications. PEG-ADA may restore and sustain immunity for many years, but is very expensive and requires injections 1-2 times per week on an ongoing basis. This clinical trial is evaluating the efficacy and safety of an alternative approach, by adding a normal copy of the human ADA gene into stem cells from the bone marrow of patients with ADA-deficient SCID. Eligible patients with ADA-deficient SCID, lacking a matched sibling donor, will be eligible if they meet entry criteria for adequate organ function and absence of active infections and following the informed consent process. Bone marrow will be collected from the back of the pelvis from the patients and processed in the laboratory to isolate the stem cells and add the human ADA gene using a retroviral vector. The patients will receive a moderate dosage of busulfan, a chemotherapy agent that eliminates some of the bone marrow stem cells in the patient, to "make space" for the gene-corrected stem cells to grow once they are given back by IV. Patients will be followed for two years to assess the potentially beneficial effects of the procedure on the function of their immune system and to assess possible side-effects. This gene transfer approach may provide a better and safer alternative for treatment of patients with ADA-deficient SCID.

DETAILED DESCRIPTION:
The proposed study population is affected with adenosine deaminase-deficient severe combined immune deficiency (ADA-SCID), an autosomal recessive congenital immune deficiency. The basis of the proposed study (and product) is retroviral-mediated transduction of autologous, bone marrow derived CD34+ hematopoietic progenitor cells with the MND-ADA retroviral vector in a 5 day cell processing period. Transduction is followed by infusion of the washed cells into subjects not receiving enzyme replacement therapy with Polyethylene-conjugated ADA (PEG-ADA, ADAGEN7) who have had their PEG-ADA injections discontinued, and have undergone bone marrow cytoreductive therapy with a single non-ablative treatment course of Busulfan. The dose of cells infused will be determined by the patient-to-patient variation of the number of progenitors available from individual patients. Statistical analyses post-infusion will help determine the dose-response of the number of cells infused to the level of engraftment and resulting level of immune reconstitution. Following cellular infusion, a primary clinical end-point will be the absolute numbers of T and B lymphocytes containing the transduced ADA gene by quantitative, real-time PCR analyses. Measurement of blood mononuclear cell ADA enzyme levels will be analyzed. Based on the degree of marking of lymphocytes and of granulocytes, the selective advantage of lymphocytes may be gauged. Subjects will be monitored for the development of clonal proliferation, under the 15 year plan required by the FDA. One major aim of the study will be to see if subjects can remain off PEG-ADA and maintain protective immunity from the population of transduced lymphocytes arising from transduced progenitors. If sufficient gene-modified cells result, and PEG-ADA enzyme replacement therapy can be permanently discontinued, the advantage of this therapeutic approach may change the standard of care for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Children > 1.0 months of age with a diagnosis of ADA-deficient SCID based on:

   * Confirmed absence (<3% of normal levels) of ADA enzymatic activity in peripheral blood or (for neonates) umbilical cord erythrocytes and/or leukocytes, or in cultured fetal cells derived from either chorionic villus biopsy or amniocentesis, prior to institution of enzyme replacement therapy.

   AND
   * Evidence of severe combined immunodeficiency based on either:

     * Family history of first order relative with ADA deficiency and clinical and laboratory evidence of severe immunologic deficiency,

   OR
   * Evidence of severe immunologic deficiency in subject based on lymphopenia (absolute lymphocyte count <200) or severely decreased T lymphocyte blastogenic responses to phytohemagglutinin (deltaCPM<5,000), prior to institution of immune restorative therapy.

   OR
   * Fulfillment of criterion:

     * A in addition to evidence of genetic mutations affecting the ADA gene as determined by a CLIA certified laboratory and clinical evidence of combined immunodeficiency based on lymphopenia (absolute lymphocyte counts <2SD of age-matched control values) and hypogammaglobulinemia (<2SD of age-matched control values) or lack of specific antibody response to vaccination. In addition, for patients to be eligible under this criterion, they must present with a clinical history indicating life-threatening illness characterized by increased frequency and/or severity of infections resulting in hospitalization and/or the administration of intravenous antibiotics, for bacterial or opportunistic infection.
2. Ineligible for allogeneic (matched sibling) bone marrow transplantation (BMT):

   * Absence of a medically eligible HLA-identical sibling with normal immune function who may serve as an allogeneic bone marrow donor.
3. Written informed consent according to guidelines of the Institutional Review Board (IRB) at the University of California Los Angeles (UCLA).

This study is also open to delayed/late onset ADA-deficient patients who fulfill the criteria 1, 2.A, and 3 and who are not receiving PEG-ADA treatment after being invited to discuss all alternative treatment options with a physician not connected with the protocol.

Exclusion Criteria:

1. Age less than 1 month
2. Hematologic

   a. Anemia (hemoglobin <10.5 mg/dl at <2 years of age, or < 11.5 at >2 years of age,with normal serum iron studies). b. Neutropenia i. absolute granulocyte count <500/mm3 or ii. absolute granulocyte count 500-999/mm3 (1 month - 1 year of age) or 500-1499/mm3 (> 1 year of age)] and bone marrow aspirate and biopsy showing myelodysplasia or other gross abnormality. c. Thrombocytopenia (platelet count 150,000/mm3, at any age). d. PT or PTT >2X normal. e. Cytogenetic abnormalities on peripheral blood, or on cells collected by amniocentesis, if diagnosed in utero.
3. Infectious

   a. Evidence of active opportunistic infection or infection with HIV-1, hepatitis B, CMV or parvovirus B 19 by DNA PCR at time of assessment.
4. Pulmonary

   1. Resting O2 saturation by pulse oximetry <95%.
   2. Chest x-ray indicating active or progressive pulmonary disease.
5. Cardiac

   1. Abnormal electrocardiogram (EKG) indicating cardiac pathology.
   2. Uncorrected congenital cardiac malformation.
   3. Active cardiac disease, including clinical evidence of congestive heart failure,cyanosis, hypotension.
6. Neurologic

   1. Significant neurologic abnormality by examination.
   2. Uncontrolled seizure disorder.
7. Renal

   1. Renal insufficiency: serum creatinine > or = 1.2 mg/dl, or > or = 3+ proteinuria.
   2. Abnormal serum sodium, potassium, calcium, magnesium, phosphate at grade III or IV by Division of AIDS Toxicity Scale.
8. Hepatic/GI:

   1. Serum transaminases > 5X normal.
   2. Serum bilirubin > 3.0 mg/dl.
   3. Serum glucose > 250mg/dl.
   4. Intractable severe diarrhea.
9. Oncologic (see below*)

   1. Evidence of active malignant disease other than dermatofibrosarcoma protuberans (DFSP)
   2. Evidence of DFSP expected to require anti-neoplastic therapy within the 5 years following the infusion of genetically corrected cells
   3. Evidence of DFSP expected to be life limiting within the 5 years following the infusion of genetically corrected cells
10. Known sensitivity to Busulfan
11. General

    1. Expected survival <6 months.
    2. Pregnant.
    3. Major congenital anomaly.
    4. Medically eligible HLA-matched sibling.
    5. Other conditions which in the opinion of the P.I. or co-investigators, contra-indicate infusion of transduced cells or indicate patient's inability to follow protocol.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald B. Kohn, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Candotti F, Shaw KL, Muul L, Carbonaro D, Sokolic R, Choi C, Schurman SH, Garabedian E, Kesserwan C, Jagadeesh GJ, Fu PY, Gschweng E, Cooper A, Tisdale JF, Weinberg KI, Crooks GM, Kapoor N, Shah A, Abdel-Azim H, Yu XJ, Smogorzewska M, Wayne AS, Rosenblatt HM, Davis CM, Hanson C, Rishi RG, Wang X, Gjertson D, Yang OO, Balamurugan A, Bauer G, Ireland JA, Engel BC, Podsakoff GM, Hershfield MS, Blaese RM, Parkman R, Kohn DB. Gene therapy for adenosine deaminase-deficient severe combined immune deficiency: clinical comparison of retroviral vectors and treatment plans. Blood. 2012 Nov 1;120(18):3635-46. doi: 10.1182/blood-2012-02-400937. Epub 2012 Sep 11. PMID 22968453
- [Derived] White SL, Lee TD, Toy T, Carroll JE, Polsky L, Campo Fernandez B, Davila A, Kohn DB, Chang VY. Evaluation of clonal hematopoiesis in pediatric ADA-SCID gene therapy participants. Blood Adv. 2022 Nov 8;6(21):5732-5736. doi: 10.1182/bloodadvances.2022007803. PMID 35914227
- [Derived] Reinhardt B, Habib O, Shaw KL, Garabedian E, Carbonaro-Sarracino DA, Terrazas D, Fernandez BC, De Oliveira S, Moore TB, Ikeda AK, Engel BC, Podsakoff GM, Hollis RP, Fernandes A, Jackson C, Shupien S, Mishra S, Davila A, Mottahedeh J, Vitomirov A, Meng W, Rosenfeld AM, Roche AM, Hokama P, Reddy S, Everett J, Wang X, Luning Prak ET, Cornetta K, Hershfield MS, Sokolic R, De Ravin SS, Malech HL, Bushman FD, Candotti F, Kohn DB. Long-term outcomes after gene therapy for adenosine deaminase severe combined immune deficiency. Blood. 2021 Oct 14;138(15):1304-1316. doi: 10.1182/blood.2020010260. PMID 33974038
- [Derived] Shaw KL, Garabedian E, Mishra S, Barman P, Davila A, Carbonaro D, Shupien S, Silvin C, Geiger S, Nowicki B, Smogorzewska EM, Brown B, Wang X, de Oliveira S, Choi Y, Ikeda A, Terrazas D, Fu PY, Yu A, Fernandez BC, Cooper AR, Engel B, Podsakoff G, Balamurugan A, Anderson S, Muul L, Jagadeesh GJ, Kapoor N, Tse J, Moore TB, Purdy K, Rishi R, Mohan K, Skoda-Smith S, Buchbinder D, Abraham RS, Scharenberg A, Yang OO, Cornetta K, Gjertson D, Hershfield M, Sokolic R, Candotti F, Kohn DB. Clinical efficacy of gene-modified stem cells in adenosine deaminase-deficient immunodeficiency. J Clin Invest. 2017 May 1;127(5):1689-1699. doi: 10.1172/JCI90367. Epub 2017 Mar 27. PMID 28346229

RESULTS

PARTICIPANT FLOW:
Groups:
- Gamma-retroviral-mediated ADA Gene Transfer: Transfer of the human ADA gene to isolated CD34+ cells from the bone marrow.
  ADA gene transfer: Autologous CD34+ cells transduced with the gamma-retroviral vector, MND-ADA, carrying the human ADA gene.
Period: Overall Study
Arm/Group | Gamma-retroviral-mediated ADA Gene Transfer
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Pre-treatment
Groups:
- Experimental Retroviral-mediated ADA Gene Transfer: Transfer of the human ADA gene to isolated CD34+ cells from the bone marrow
Arm/Group | Experimental Retroviral-mediated ADA Gene Transfer
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Examine the safety of the procedure: harvesting bone marrow, isolating CD34+ hematopoietic stem/progenitor cells, performing ex vivo gene transduction with the MND-ADA gamma-retroviral vector, giving 90 mg/m2 busulfan to "make space" in the bone marrow to aid engraftment, and re-infusing the autologous gene-modified cells.
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- Gamma-retroviral Mediated ADA Gene Transfer: Transfer of the human ADA gene to isolated CD34+ cells from the bone marrow
Arm/Group | Gamma-retroviral Mediated ADA Gene Transfer
Number analyzed (Participants) | 10
participants
  Expected Grade 3 or 4 AE related to procedure | 10
  Unexpected Grade 3 or 4 AE related to procedure | 9
  Grade 3 or 4 AE related to study product | 0
  Alive | 10
  Deaths | 0

2. Secondary Outcome: Number of Participants With Greater Than 1% of Gene-Modified Cells in the Peripheral Blood
Description: As measured by quantitative polymerase chain reaction in peripheral blood cells separated into mononuclear and granulocyte fractions.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Gamma-retroviral Mediated ADA Gene Transfer
Number analyzed (Participants) | 10
participants
  For peripheral blood mononuclear cells | 10
  for peripheral blood granulocytes | 4

3. Secondary Outcome: Number of Participants Reaching the Normal Range of ADA Enzyme Activity
Description: As measured by ADA enzyme activity in peripheral blood mononuclear cells
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Gamma-retroviral Mediated ADA Gene Transfer
Number analyzed (Participants) | 10
participants | 9

ADVERSE EVENTS:
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 18, 21, 24 months
Arm/Group | Retroviral-mediated ADA Gene Transfer
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retroviral-mediated ADA Gene Transfer (N=10)
Infection requiring hospitalization (Immune system disorders) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Retroviral-mediated ADA Gene Transfer (N=10)
neutropenia (Blood and lymphatic system disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No